CLINICAL TRIAL: NCT04649190
Title: Post-TAVI Coronary Access Study
Acronym: PTCA
Status: Completed | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Issi Barbash, Prof, Sheba Medical Center
Other Study IDs: SHEBA-13-0685-IB-CTIL-B
Record Dates: First submitted 2020-11-24; First posted 2020-12-02 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TAVI
  Interventions: Device: TAVI

INTERVENTIONS:
Device: TAVI — Coronary access for PCI after TAVI

SUMMARY:
Coronary access after trans-catheter aortic valve implantation (TAVI) remains a major challenge. With the evolution of TAVI procedure and the inclusion of lower-risk patients with aortic stenosis, future coronary access is an even greater concern, because this lower-risk patient group has a greater cumulative risk of requiring coronary angiography for acute coronary events compared to their octogenarian counterparts.

It is only speculated that the intra-annular position of the self-expandable valves together with the frame covering coronary ostia would impose a significant technical challenge as compared to the balloon-expandable valve (1). However, this remains to be proven. With any valve used, increased catheter manipulations may result in longer fluoroscopy times, larger volumes of contrast, and reduced imaging quality due to non-selective injections (2).

Although complex, coronary procedures after TAVR are considered relatively safe and feasible on experience hands (3-6). A number of techniques to increase the likelihood of successful coronary intubation after TAVR have been described in the published reports and include the use of intracoronary guidewires (1), as well as balloon-assisted tracking with guideliner extension (7). It is therefore essential to fully understand the potential challenges of coronary angiography and PCI in this specific patient population. Guidance by a specific algorithm may help to overcome difficulties in coronary angiography and facilitate selective coronary intubation particularly during primary PCI (8).

ELIGIBILITY:
Inclusion Criteria:

1. Prior TAVI for aortic stenosis or regurgitation in bicuspid or tricuspid valve
2. Clinical indication for PCI

Exclusion Criteria:

1. Prior TAVI valve-in-valve procedures
2. Prior TAVI-in-TAVI procedures

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects who underwent TAVI at any time point prior to index PCI procedure, and who have clinical indication for PCI will be included in the present study. Consecutive subjects of both genders will be enrolled at various sites in Europe, United States and Asia (See Appendix 1). The study procedures, clinical management and follow up will be done at each participating center.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
PCI device success | 5 year

SECONDARY OUTCOMES:
Successful delivery, balloon expansion, and deployment of the first assigned device, at the intended target lesion | 5 year
Successful withdrawal of the device delivery system | 5 year
Attainment of a final in-stent or in-scaffold residual stenosis of <20% | 5 year
Final TIMI flow | 5 year
Successful selective engagement of guiding catheter | 5 year
Incidence of procedural complications | 5 year
Procedural mortality | 5 year

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No